CLINICAL TRIAL: NCT06500143
Title: The RESIDUAL Study : Residual Gastric Content After Holding of Glucagon-like Peptide-1 Receptor Agonists Before Elective Surgery: a Cross-sectional Study
Brief Title: Residual Gastric Content After Holding of Glucagon-like Peptide-1 Receptor Agonists Before Elective Surgery
Acronym: RESIDUAL
Status: Completed | Type: Observational
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Institut de Cardiologie de Montréal (Unknown)
Responsible Party: Sponsor
Other Study IDs: MP-12-2025-3794
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Gastric Retention
Keywords: glucagon-like peptide 1; gastric ultrasound; surgery; diabetes; weight loss; increased residual gastric content; semaglutide; dulaglutide
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLP-1RA agonists users: Participants presenting for elective surgery and taking once-weekly semaglutide or dulaglutide as part of their usual treatment with the last dose at least 7 days before surgery
  Interventions: Diagnostic Test: Gastric ultrasound
- Control group: Participants presenting for elective surgery and not taking semaglutide or dulaglutide
  Interventions: Diagnostic Test: Gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric ultrasound — Using a curved array low-frequency abdominal probe (2-5 MHz) with abdominal presets and with the patient in right lateral decubitus position, the gastric antrum will be identified in a standardized plane at the level of the aorta. The stomach will be considered empty if the antrum appears flat or round with anterior and posterior walls collapsed. Normal gastric secretions and clear fluids have an anechoic or hypoechoic aspect on ultrasonography. Solid or thick fluids have a hyperechoic aspect and can create "ring-down" artifacts blurring gastric content, its posterior wall, the pancreas and the aorta. Following qualitative examination, quantitative assessment will be performed if there is presence of clear fluids. The cross-sectional area (CSA) of the antrum will be measured with three measurements to calculate a mean value.

SUMMARY:
Glucagon-like peptide-1 agonists (GLP-1RA) are a family of medications used for diabetes and weight loss. One of their effect is to slow down stomach emptying. The goal of this study is to evaluate the effect of GLP-1RA on the effectiveness of fasting before a scheduled surgery.

The question it aims to answer is: does this kind of medication increase the risk of having food or too much liquid in the stomach before a scheduled surgery, even if the minimum 6 hour fast is done?

For this project, researchers will use gastric ultrasound to compare participants already taking one of these medications as part of their home treatment to participants who are not taking them. Gastric ultrasound is a simple bedside exam using an echography machine that takes less than 5 minutes to do.

Participants will:

-Have a gastric ultrasound performed on them before their surgery

DETAILED DESCRIPTION:
Background: Glucagon-like peptide-1 receptor agonists (GLP-1RA) are glucose-lowering drugs that act through three mechanisms: stimulation of insulin secretion, inhibition of glucagon secretion and decrease of gastric emptying. The GLP-1RA are now an important part of glycemic control in type 2 diabetes mellitus (T2DM). Recently, GLP-1 RA have received approval for weight loss, expanding their use in overweight or obese non-diabetic patients.The effect of GLP-1RA on decreased gastric emptying has long been established but he clinical implication of this in the periprocedural setting is uncertain. Recent guidelines recommend holding the weekly-dosed for at least a week before elective surgery. Considering the extended half-lives of once-weekly GLP-1RA (approximately 6 days for semaglutide and 5 days for dulaglutide), it is unclear if following those guidelines is sufficient to make sure patients are not at high risk of aspiration

Hypothesis: This study will compare ultrasound-assessed residual gastric content (RGC) between once-weekly GLP-1RA users that stopped their medication for 7 days or more before elective surgery and patients not taking GLP-1RA. The investigators hypothesized that even with appropriate holding of GLP-1RA, those patients may have increased RGC and be at higher risk of aspiration.

Objectives:

Primary objective:

• To investigate the relation between GLP-1RA use and increased RGC

Secondary objectives:

* To assess the relation between the number of days since the last dose of GLP-1RA and increased RGC
* To assess the relation between the dose of GLP-1RA and RGC

Exploratory objectives:

* To explore the relation between other known risk factors of gastroparesis and increased RGC
* To explore the relation between the time since the last oral intake and increased RGC

Methods : A gastric ultrasound (GUS)will be performed on all patients to assess RGC using a published validated and reproductible method used in recent trials. The acquisition of images will be performed by a blinded anesthesiologist or anesthesiology resident using a dedicated ultrasound machine. The images will be saved and reviewed by another blinded trained anesthesiologist.

Significance/importance: The results of this study could challenge the actual recommendations for GLP-1RA stoppage before surgery and help improve perioperative care for patients taking GLP-1RA.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class 1-4 patients
* Age ≥ 18 years old
* Fasted state (2 hours for clear liquids, 6 hours for solids)
* Elective surgery
* Last dose of once-weekly semaglutide or dulaglutide 7 days or more before surgery (for GLP-1RA group)

Exclusion Criteria:

* Last dose of GLP-1RA less than 7 days before surgery
* Inability to lay on the right-side for ultrasound
* Pregnancy
* History of gastric surgery or large hiatal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult population undergoing elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Increased residual gastric content | Preoperative (day of surgery)
  The primary endpoint will be the prevalence of increased residual gastric content defined by the presence of any of the following:
  * Solid or thick fluid content on gastric ultrasound
  * Content of more than 1.5 mL/kg of clear fluids on gastric ultrasound using the following formula : Gastric volume (mL) = 27 + [14.6 × right lateral cross-sectional area (in cm2)] - [1.28 × age (in years)]

CONTACTS AND LOCATIONS:
Overall Officials: Louis Morisson, MD, MSc, Principal Investigator — CIUSS de l'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada